CLINICAL TRIAL: NCT04582942
Title: Improved Bowel Preparation Method for Colonoscopy Based on Different Risk Stratification：a Multicenter, Endoscopist-blinded Randomized Controlled Trial
Brief Title: Improved Bowel Preparation Method for Colonoscopy Based on Different Risk Stratification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan Central Hospital (Other); Wuhan Third Hospital (Other); The General Hospital of Central Theater Command (Other); The Third People's Hospital of Hubei Province (Other); Wuhan Puren Hospital (Other); Wuhan Puai Hospital (Unknown); Tian You Hospital Affiliated to Wuhan University of Science and Technology (Unknown); Wuhan Red Cross Hospital (Unknown)
Responsible Party: Principal Investigator, ChenMingkai, Chief physician of Department of Gastroenterology I, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2019-X2-73
Record Dates: First submitted 2020-09-25; First posted 2020-10-12 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Bowel Preparation Before Colonoscopy
Keywords: Colonoscopy; Lactulose; Polyethylene glycol; Bowel preparation
MeSH Terms: interventions — Lactulose

STUDY DESIGN:
Intervention Model Description: Patients scheduled for colonoscopy were stratified into low- and high-risk patients based on the inclusion criteria. Low- and high-risk patients were randomized to the PEG alone or lactulose combined with PEG group respectively.
Who Masked: Investigator
Masking Description: The allocation assignment of patients was performed by a designated technician at each center based on a computer-generated random sequence. The designated technician was not involved in the colonoscopy procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG (low-risk patients and high-risk patients) (Placebo Comparator): The dosing regimen of low-risk patients and high-risk patients will only be PEG.
  Interventions: Drug: PEG
- PEG+lactulose (low-risk patients and high-risk patients) (Experimental): The dosing regimen of low-risk patients and high-risk patients will be PEG combined with lactulose.
  Interventions: Drug: PEG+lactulose

INTERVENTIONS:
Drug: PEG — Patients began to drink 1 L of PEG at 8:00 PM on the day before colonoscopy at a rate of 250 mL every 10- 15 minutes. On the day of the procedure, patients took the remaining 2 L of PEG 4-6 hours before colonoscopy.
  Other Names: only used PEG
  Arms: PEG (low-risk patients and high-risk patients)
Drug: PEG+lactulose — On the day before colonoscopy , Patients took 45 mL lactulose solution at 7:00 PM. And then Patients began to drink 1 L of PEG at 8:00 PM at a rate of 250 mL every 10- 15 minutes. On the day of the procedure, patients took 45 mL lactulose solution and the remaining 2 L of PEG 4-6 hours before colonoscopy.
  Other Names: PEG combined with lactulose
  Arms: PEG+lactulose (low-risk patients and high-risk patients)

SUMMARY:
The purpose of this study is to evaluate the efficacy of polyethylene glycol（PEG） combined with lactulose for bowel preparation before colonoscopy in low-risk patients and high-risk patients.

DETAILED DESCRIPTION:
The quality of bowel preparation is crucial for colonoscopy. Some high-risk factors for inadequate bowel preparation have been identified , including age >70, previous colon surgery, constipation, diabetes, Parkinson's disease, history of stroke or spinal cord injury, prior history of inadequate bowel preparation, body mass index (BMI) >25, use of tricyclic antidepressant or narcotics. Patients were considered as high risk if they have any of the above factors and considered as low risk if they did not have any of these risk factors.This is a multicenter, endoscopist-blinded study to compare the efficacy of PEG combined with lactulose and PEG alone in bowel preparation. In colonoscopy procedures, endoscopists who were blinded to the intervention evaluated the overall quality of colonoscopy cleaning according to the Boston Bowel Preparation Scale. Patients' tolerance, defecation, adverse events and adenoma detection rate (ADR) were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Adults undergoing colonoscopy.

Exclusion Criteria:

* 1.presence of any contraindications for colonoscopy (gastrointestinal obstruction or perforation,severe acute inflammatory bowel disease,toxic megacolon,severe heart failure,unable to swallow,severe heart failure,etc);
* 2.Patients with galactosemia;
* 3. hypersensitivity to any of the ingredients;
* 4.Pregnancy or lactation;
* 5.Use of lactulose,prokinetic agents or purgatives within 7 days;
* 6.Unwilling to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2028 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | during colonoscopy
  Cleanliness of the colon during colonoscopy will be evaluated by the Boston Bowel Preparation Scale which is a 4-point scoring system applied to each of 3 broad regions of the colon: the right side, the transverse section, and the left side. The total BBPS score ranged from 0 to 9. If total BostonBowel Preparation Score ≥6 with each segmental BBPS≥2, we regard it as adequate bowel preparation.

SECONDARY OUTCOMES:
Adenoma Detection Rate | 2 days
  Diagnosis was confirmed by histologic examination
Rate of adverse events | 2 days
  adverse events, such as vomiting, nausea, headache, abdominal distention,abdominal pain.
Cecal intubation rate | during colonoscopy
  Colonoscopy reaches cecal region.
Cecal intubation time | during colonoscopy
  Colonoscopy reaches cecal region.
Withdrawal time | during colonoscopy
  The time from the cecum to the anus, but excluded time for biopsy performance or removal of polyps.
defecation frequency | 2 days
  Frequency of bowel movement.
Willingness to repeat bowel preparation | 2 days
  The number of patients have a willingness to undergo a repeated bowel preparation if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, M.D, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Bai Y, Fang J, Zhao SB, Wang D, Li YQ, Shi RH, Sun ZQ, Sun MJ, Ji F, Si JM, Li ZS. Impact of preprocedure simethicone on adenoma detection rate during colonoscopy: a multicenter, endoscopist-blinded randomized controlled trial. Endoscopy. 2018 Feb;50(2):128-136. doi: 10.1055/s-0043-119213. Epub 2017 Oct 6. PMID 28985630
- [Background] Kang X, Zhao L, Zhu Z, Leung F, Wang L, Wang X, Luo H, Zhang L, Dong T, Li P, Chen Z, Ren G, Jia H, Guo X, Pan Y, Guo X, Fan D. Same-Day Single Dose of 2 Liter Polyethylene Glycol is Not Inferior to The Standard Bowel Preparation Regimen in Low-Risk Patients: A Randomized, Controlled Trial. Am J Gastroenterol. 2018 Apr;113(4):601-610. doi: 10.1038/ajg.2018.25. Epub 2018 Mar 13. PMID 29533397
- [Background] Lu J, Cao Q, Wang X, Pu J, Peng X. Application of Oral Lactulose in Combination With Polyethylene Glycol Electrolyte Powder for Colonoscopy Bowel Preparation in Patients With Constipation. Am J Ther. 2016 Jul-Aug;23(4):e1020-4. doi: 10.1097/MJT.0000000000000351. PMID 26658804